CLINICAL TRIAL: NCT02090192
Title: Acute and Chronic Effects of Whole-body Vibration on Mobility, Muscle Strength, Bone and General Health Status in the Frail Elderly
Brief Title: Effects of Whole-body Vibration in the Frail Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Zhang (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, Doctor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChinaPLAGH-2013FC3009
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Sarcopenia;; Osteoporosis
Keywords: Whole-body vibration;; Frail Elderly;; Blood flow;; Bone density; Mobility;; Balance;; Muscle strength;; Lower Extremity;; Musculoskeletal System;; Health Status;; Exercise;; Mechanical Oscillation
MeSH Terms: conditions — Sarcopenia; Osteoporosis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- WBV training (Experimental): Whole-body vibration training was performed on a commercial Galileo machine (Germany). Participants were required to stand on the moveable rectangular platform and positioned their feet at an equal and standardized distance from the axis of rotation so that the vertical vibration amplitude was 1-3 mm. The frequency was set at 6-26 Hz. The vibration protocol consisted of four to five bouts (60 seconds for each bout), and three to five times a week for 12 weeks. The positions taken by the subjects differed according to their function. Participants who could stand independently were instructed to adopt a "partial squat" position with slight flexion at the hips, knees, and ankle joints to damp the vibrations approximately at the pelvic level.
  Interventions: Procedure: WBV training
- WBV+ PRT training (Experimental)
  Interventions: Procedure: WBV training; Procedure: PRT training
- PRT training (Active Comparator)
  Interventions: Procedure: PRT training
- Control group (Placebo Comparator)

INTERVENTIONS:
Procedure: WBV training
  Arms: WBV training; WBV+ PRT training
Procedure: PRT training
  Arms: PRT training; WBV+ PRT training

SUMMARY:
Objective: To study the acute and chronic effects of whole-body vibration (WBV) exercises on the lower extremity blood flow, mobility function, balance, muscle strength, bone density, and general health status, and its feasibility as an intervention in frail elderly patients.

Design: Randomized controlled trial. Subjects: The frail older persons meeting the Fried Frailty Criteria.

Interventions: All eligible subjects were randomly assigned to 4 groups:

(1) WBV group: Subjects received a whole-body vibration exercise alone; (2) Progressive resistance training (PRT) group: Subjects received progressive resistance training; (3) WBV+ PRT group: Subjects received the whole-body vibration and progressive resistance training; (4) Control group: Subjects received no intervention/training. The periods of intervention are 12 weeks.

Main measures: The lower extremities blood flow (the diameters and red blood cell velocity of the common femoral artery), timed up and go test, 30-second chair stand test, five times sit to stand test, lower extremities muscle strength, balance function, balance confidence, bone density, and general health status was assessed at the beginning of the study, at instant, 12 weeks and 24 month after the intervention.

Study hypothesis: Whole-body vibration exercise is a safe and effective method that can improve the lower extremity blood flow, mobility function, balance, muscle strength, bone density, and general health status in the frail elderly.

ELIGIBILITY:
Inclusion Criteria:

* ≥75 years old
* Fried Frailty Criteria
* Mini Mental State Examination score ≥18

Exclusion Criteria:

* Recent fractures (≤6 months)
* Gallbladder or kidney stones
* Malignancies
* Rheumatic arthritis
* Epilepsy
* Serious heart sicknesses or an implant, and bypass stent or cardiac pacemaker
* Any diseases to be associated with a life expectancy of less than 12 months

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of the common femoral artery's blood flow from Baseline to 60min post-WBV | 60min post-WBV
Change of lower extremities muscle strength from Baseline to 3 month post-WBV | 3 month post-WBV
Change of "timed up and go" test (TUGT) from Baseline to 3 month post-WBV | 3 month post-WBV
Change of 30-second chair stand test from Baseline to 3 month post-WBV | 3 month post-WBV
Change of balance function from Baseline to 3 month post-WBV | 3 month post-WBV
Change of balance confidence from Baseline to 3 month post-WBV | 3 month post-WBV
Change of bone density from Baseline to 6 month post-WBV | 6 month post-WBV
Change of general health status (SF-12 score) from Baseline to 6 month post-WBV | 6 month post-WBV

CONTACTS AND LOCATIONS:
Overall Officials: Changshui Weng, Bachelor, Study Director — Chinese PLA General Hospital
Locations (1):
- Rehabilitation Department, Nanlou, Chinese PLA general hospital, Beijing, Beijing Municipality, China